CLINICAL TRIAL: NCT02358382
Title: The Management of Systemic-Pulmonary Collateral Blood Flow in Cyanotic Children During Cardiopulmonary Bypass - Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13CC21
Record Dates: First submitted 2014-11-26; First posted 2015-02-09 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha Stat (No Intervention): Standard CPB blood gas management conditions
- pH Stat (Experimental): pH stat blood gas management conditions.
  Interventions: Drug: pH Stat

INTERVENTIONS:
Drug: pH Stat — pH stat blood gas management - increased carbon dioxide content of administered gas mixture.
  Arms: pH Stat

SUMMARY:
The purpose of the study is to determine whether it is possible to manage the flow of blood through blood vessels using varying levels of carbon dioxide during cardiac surgery, and what effect this has on how well the major organs of the body work.

DETAILED DESCRIPTION:
A great number of studies have shown that MAPCAs are a real issue for these patients, who require far higher blood flows than previously suggested. However, the optimal method of CPB is still unknown. Recent research by Sakamoto et al., showed that a raised carbon dioxide (pCO2) increased brain blood flow in cyanotic patients, suggesting a noticeable decrease in aorto-pulmonary blood shunting. However, the mechanism of this action is not understood and it is unclear if this observation is an associated or causative one. Whilst the vasoconstrictive (narrowing of vessels) effect of hypoxia has been well documented, with and without high carbon dioxide, there are no reports indicating that pCO2 alone increases the narrowing of blood vessels in the lung. We hypothesize that a rise in pCO2 could cause a shift in blood flow from pulmonary to systemic circulation, either through direct constricting action on MAPCA vessels, or through a vasoconstriction of blood vessels in the lung. Furthermore, we predict the phenomenon could potentially be used to optimize the method of treatment, ensuring that vital organs receive the correct amount of blood flow during the surgical correction of these rare congenital heart diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents/guardians are willing and able to provide written informed consent for participation in the study
* Patients undergoing elective TCPC surgery
* MRI proven presence of MAPCA vessels
* Patients between 1 day and 5 years of age

Exclusion Criteria:

* Emergency surgery
* Documented history of cognitive impairment (may have an effect on biochemical markers of cerebral injury)
* Documented history of major organ dysfunction

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
MAPCA Flow | During surgery
  To determine the optimal conditions for treating cyanotic patients with MAPCAs on CPB

SECONDARY OUTCOMES:
Maximum levels of Biochemical markers of Cerebral and Tissue Injury, as measure by Neurone-Specific Enolase, Creatine Kinase, Gamma Glutamyl Transferase, Lactate Dehydrogenase and Near Infrared Spectroscopy | 3 days Post Surgical Period
  To determine if increased pCO2 levels results in altered organ and tissue perfusion as measure by Neurone-Specific Enolase, Creatine Kinase, Gamma Glutamyl Transferase, Lactate Dehydrogenase and Near Infrared Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Issitt, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Background] Whitehead KK, Gillespie MJ, Harris MA, Fogel MA, Rome JJ. Noninvasive quantification of systemic-to-pulmonary collateral flow: a major source of inefficiency in patients with superior cavopulmonary connections. Circ Cardiovasc Imaging. 2009 Sep;2(5):405-11. doi: 10.1161/CIRCIMAGING.108.832113. Epub 2009 Jul 8. PMID 19808629
- [Background] Fujii Y, Kotani Y, Kawabata T, Ugaki S, Sakurai S, Ebishima H, Itoh H, Nakakura M, Arai S, Kasahara S, Sano S, Iwasaki T, Toda Y. The benefits of high-flow management in children with pulmonary atresia. Artif Organs. 2009 Nov;33(11):888-95. doi: 10.1111/j.1525-1594.2009.00895.x. Epub 2009 Oct 10. PMID 19817735
- [Background] Haworth SG, Macartney FJ. Growth and development of pulmonary circulation in pulmonary atresia with ventricular septal defect and major aortopulmonary collateral arteries. Br Heart J. 1980 Jul;44(1):14-24. doi: 10.1136/hrt.44.1.14. No abstract available. PMID 7426156
- [Background] Liao PK, Edwards WD, Julsrud PR, Puga FJ, Danielson GK, Feldt RH. Pulmonary blood supply in patients with pulmonary atresia and ventricular septal defect. J Am Coll Cardiol. 1985 Dec;6(6):1343-50. doi: 10.1016/s0735-1097(85)80223-0. PMID 4067114
- [Background] Baile EM, Ling H, Heyworth JR, Hogg JC, Pare PD. Bronchopulmonary anastomotic and noncoronary collateral blood flow in humans during cardiopulmonary bypass. Chest. 1985 Jun;87(6):749-54. doi: 10.1378/chest.87.6.749. PMID 3996062
- [Background] Sakamoto T, Kurosawa H, Shin'oka T, Aoki M, Isomatsu Y. The influence of pH strategy on cerebral and collateral circulation during hypothermic cardiopulmonary bypass in cyanotic patients with heart disease: results of a randomized trial and real-time monitoring. J Thorac Cardiovasc Surg. 2004 Jan;127(1):12-9. doi: 10.1016/j.jtcvs.2003.08.033. PMID 14752407
- [Background] Kato M, Staub NC. Response of small pulmonary arteries to unilobar hypoxia and hypercapnia. Circ Res. 1966 Aug;19(2):426-40. doi: 10.1161/01.res.19.2.426. No abstract available. PMID 5914855